CLINICAL TRIAL: NCT04440904
Title: Anatomical Study of Aorta Balloon Occlusion Based on CT Angiography：A Retrospective Study
Brief Title: Anatomical Study of Aorta Balloon Occlusion Based on CT Angiography
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-333
Record Dates: First submitted 2020-06-16; First posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: CT Angiography; Marker; Structural
Keywords: CT angiography; Aorta; Anatomy; Aortic balloon occlusion; Body surface markers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Characteristic of aortic length and body surface mark: The diameters and lengths of blood vessels and the distances on the body surface were measured by three-dimensional reconstruction using related Software on CT Workstation
  Interventions: Device: CT workstation (Syngo Via VB10B, Siemens, Germany)

INTERVENTIONS:
Device: CT workstation (Syngo Via VB10B, Siemens, Germany) — Multiplanar reconstruction, curvature plane reconstruction, and volume rendering were used for three-dimensional reconstruction to measure the diameters and lengths of blood vessels and the distances on the body surface

SUMMARY:
Aortic balloon occlusion can be used by emergency physicians to rescue patients with massive bleeding.The purpose of this study is to study the anatomical characteristics of aortic balloon occlusion based on aortic CT angiography, so as to provide evidence for improving the success rate of aortic balloon occlusion guided by body surface markers.

DETAILED DESCRIPTION:
Study Design:

This study is a retrospective descriptive study. The study will be conducted by Radiology Department, Second Affiliated Hospital, Zhejiang University.

Selection of patients:

The investigators included 57 patients who underwent enhanced contrast full-length aortic CTA scanning in the Radiology Department of Grade 3A General Hospital affiliated to a university from April to December 2019. Data of all participants following no apparent vascular tortuosity in CT diagnosis aged 18-70 years with contrast-enhanced computed tomography (CT) images of chest, abdomen, and pelvis from April to December in 2019 were analyzed. Participants whose images accompanied by vascular malformation, poor contrast enhancement, and history of aortic surgery were precluded.

Method General data of patients were collected through the hospital's electronic medical record system, including age, sex, height, weight, average body mass index ((Body Mass Index,BMI), history of surgery, etc.

The CTA examination of the participants' full aorta was performed with a 128-slice dual-energy CT scanner (Siemens, Germany), and the images were saved in the database. After screening the suitable participants, the images were transmitted to the CT workstation (Syngo VB10B Image processing system, Siemens, Germany). Multiplanar reconstruction, curvature plane reconstruction, and volume rendering were used for three-dimensional reconstruction. The diameters and lengths of blood vessels and the distances on the body surface were measured. The diameters of blood vessels included the diameter of the aorta at the edge of left subclavian artery, celiac trunk, lowest renal artery, and aortic bifurcation. The intravascular length included the lengths of zone I, zone II, zone III and the descending aorta. The length from the bilateral femoral artery puncture site to the midpoint of zone I and III, left subclavian artery, celiac trunk, lowest renal artery and aortic bifurcation, and the distances on the body surface included the distance from the bilateral femoral artery puncture site to the suprasternal notch, xiphoid process and umbilicus.

The results were described as mean ±standard deviation. SPSS20.0 software (IBM, USA) was used for analysis. Paired sample t-test was used to compare the differences between the left and right sides of the data. The difference was statistically significant when the P value was less than 0.05.

Data Management and Confidentiality Data Management: Using paper version for data management and storage. The person responsible for collecting paper version will input data in Excel database, summary paper and electronic versions for further statistical analysis and preservation.

Security measures: All records related to the identity of participants are to be confidential and not open to the public outside the scope of relevant laws or regulations.

Informed consent: This study is a retrospective study. Retrospective measurement of participants' previous aortic CTA imaging data does not infringe upon the interests of participants, so informed consent can be exempted.

Possible risks of participating in this study: disclosure of personal information.

Precautions against possible risks:

1. All the experimental data of the paper version and the electronic version shall be kept by the person in charge of the test data.
2. Close the measurement software in time after the end of the study, and confirm that the personal information has been cleared.

Intervention measures for possible risks:

If there is a disclosure of personal information, it is necessary to record the research report form and inform the person in charge of the research to intervene in time, and notify the Ethics Committee immediately.

ELIGIBILITY:
Inclusion Criteria:

* Complete full-length CTA scan of aorta
* Aged 18-70 years old
* No obvious tortuosity diagnosed by CT

Exclusion Criteria:

* Aortic dissection
* Aortic aneurysm
* Severe aortic malformation
* Severe aortic plaque
* History of aortic operation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We conduct an observational retrospective study.The patients underwent aortic CT angiography examination in the radiology department of the hospital from April to December in 2019.
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
The length from the bilateral femoral artery puncture site to the left subclavian artery, celiac trunk, lowest renal artery and aortic bifurcation | within 24 hours
  The lengths of the blood vessels were measured along the centerline of the blood vessels by multiplanar reconstruction and curvature plane reconstruction
The distances on the body surface from the bilateral femoral artery puncture site to the suprasternal notch, xiphoid process and umbilicus | within 24 hours
  The distances between the body surface mark were measured by using volume-rendering reconstruction

SECONDARY OUTCOMES:
the length of zone I | within 24 hours
  defined as the distance from the left subclavian artery to the celiac trunk
the length of zone II | within 24 hours
  defined as the distance from the celiac trunk to the lowest renal artery
the length of zone III | within 24 hours
  defined as the distance from the lowest renal artery to the aortic bifurcation

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, Zhejiang University School of Medicine & Institute of Emergency Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] White JM, Cannon JW, Stannard A, Markov NP, Spencer JR, Rasmussen TE. Endovascular balloon occlusion of the aorta is superior to resuscitative thoracotomy with aortic clamping in a porcine model of hemorrhagic shock. Surgery. 2011 Sep;150(3):400-9. doi: 10.1016/j.surg.2011.06.010. PMID 21878225
- [Background] Stannard A, Eliason JL, Rasmussen TE. Resuscitative endovascular balloon occlusion of the aorta (REBOA) as an adjunct for hemorrhagic shock. J Trauma. 2011 Dec;71(6):1869-72. doi: 10.1097/TA.0b013e31823fe90c. No abstract available. PMID 22182896
- [Background] Linnebur M, Inaba K, Haltmeier T, Rasmussen TE, Smith J, Mendelsberg R, Grabo D, Demetriades D. Emergent non-image-guided resuscitative endovascular balloon occlusion of the aorta (REBOA) catheter placement: A cadaver-based study. J Trauma Acute Care Surg. 2016 Sep;81(3):453-7. doi: 10.1097/TA.0000000000001106. PMID 27192466
- [Background] Okada Y, Narumiya H, Ishi W, Iiduka R. Anatomical landmarks for safely implementing resuscitative balloon occlusion of the aorta (REBOA) in zone 1 without fluoroscopy. Scand J Trauma Resusc Emerg Med. 2017 Jul 3;25(1):63. doi: 10.1186/s13049-017-0411-z. PMID 28673353
- [Background] Eliason JL, Derstine BA, Horbal SR, Wang NC, Holcombe SA, Chiu CH, Ross BE, Bromwell B, Morrison J, Wang SC. Computed tomography correlation of skeletal landmarks and vascular anatomy in civilian adult trauma patients: Implications for resuscitative endovascular balloon occlusion of the aorta. J Trauma Acute Care Surg. 2019 Jul;87(1S Suppl 1):S138-S145. doi: 10.1097/TA.0000000000002247. PMID 31246918